CLINICAL TRIAL: NCT04863859
Title: Persons With Dementia and Their Extended Family Caregivers: Service Use, Barriers and Needs
Brief Title: Persons With Dementia and Their Extended Family Caregivers
Acronym: CareEx
Status: Recruiting | Type: Observational
Sponsor: Karen Roberto (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Karen Roberto, University Distinguished Professor, Virginia Polytechnic Institute and State University
Organization: Virginia Polytechnic Institute and State University (Other)
Other Study IDs: 20-742; R01AG069818 (NIH)
Record Dates: First submitted 2021-04-22; First posted 2021-04-28 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Dementia; Dementia Alzheimers; Neuro-Degenerative Disease; Dementia of Alzheimer Type; Dementia Severe
Keywords: caregiving, persons living with dementia, community-based services
MeSH Terms: conditions — Dementia; Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Grandchildren: Granddaughter or Grandson of the person living with dementia who serves as the primary caregiver
- Siblings: Brother, sister, brother-in-law or sister-in-law of the person living with dementia who serves as the primary caregiver
- Nieces/Nephews: Niece or nephew of the person living with dementia who serves as the primary caregiver
- Step-Kin: Step-kin (step-daughter, step-son, step-sister, step-brother or other step-kin) of the person living with dementia who serves as the primary caregiver
- Adult Child: Adult child (son or daughter) of the person living with dementia who serves as the primary caregiver
- Spouse: Spouse (husband or wife) of the person living with dementia who serves as the primary caregiver

SUMMARY:
Immediate family members shoulder the majority of care responsibilities for persons living with dementia. However, due to various societal changes, elder care responsibilities have expanded to extended family members, including grandchildren, siblings, nieces/nephews, siblings, and step-kin.

The main objective of this study is to understand the caregiving journeys of various extended family members involved in dementia care. We aim to learn about caregivers' care management strategies; their use of home and community-based services and informal support; and barriers to service usage. We will use the results from the study to help enhance service delivery, alleviate care-related stress, and improve the quality of life of dementia patients and their caregivers.

We will use a mixed-methods design to explore the challenges faced by caregivers as well as their service usage for the person living with dementia. Our methodology involves an initial telephone interview (approx. 70 minutes) that includes open-ended questions, standard items, and structured measures, followed by an 8-day semi-structured daily diary interview about daily care responsibilities and experiences with services (15-20 minutes each evening). This study will be conducted with 240 extended family members serving as one of the main caregivers for a person living with dementia in a community setting.

ELIGIBILITY:
Inclusion Criteria:

* Speaks/reads English
* Resident of Virginia, North Carolina, Maryland, West Virginia, Tennessee, Kentucky or Washington, D.C.
* Age 18+
* Is either the grandchild, sibling, niece/nephew, step-kin, adult child or spouse of the person living with dementia
* Is providing hands-on care and/or overall management of care for a person living with dementia in the community
* Caregiver co-resides with the person with dementia or has face-to-face contact with the person with dementia at least 3 days/week
* Has no difficulty talking/hearing on the telephone

Exclusion Criteria:

* Caregiver of persons with mild cognitive impairment
* Person with dementia lives in service-enriched housing such as a continuing care community, or residential facilities, such as assisted living facilities or nursing homes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population includes extended family caregivers defined as grandchildren, siblings, nieces/nephews and step-kin of persons living with dementia. Caregivers must be as least 18 years of age and primarily responsible for the hands-on care and/or overall management of care for a person living with dementia living in the community. The study will recruit 60 grandchildren, 60 siblings, 60 nieces/nephews and 60 step-kin care givers; in additional 60 adult child and 60 spouse caregivers will be recruited for comparison purposes.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2021-09-11 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Well-Being of Person Living with Dementia | Day 1 to Day 8
  The caregiver (CG) will be asked to indicate who helped the person living with dementia (PLwD) each of the daily diary days with personal activities of daily living and instrumental activities of daily living for which they need help. CG will also be asked if there were any activities for which the PLwD needed help that day but did not receive it because no one was there to help them (PLwD Unmet Need), or they delayed receiving help or received partial help because no one was available to help them when needed (PLwD Under-met Need).
Well-Being of Caregiver: Role overload | Baseline
  Role overload, a 3-item scale will assess CG subjective appraisal of the time and effort they make in providing care. Participants rate their responses on a 4-point scale ("not at all" to "completely"). Summary scores range from 0 to 9, higher scores indicate greater role overload.
Well-Being of Caregiver: Role Captivity | Baseline
  Role captivity, a 3-item scale that assesses CG feelings that their involvement exceeds what they are willing to provide. Participants rate their responses on a 4-point scale ("not at all" to "very much"). Summary scores range from 0 to 9, higher scores indicate greater role captivity.
Well-Being of Caregiver: Work Strain | Baseline
  CG who are employed will be asked 5 work strain items that assess competing demands and strains between CG and employment outside the home. Participants rate their responses on a 4-point scale ("strongly agree" to "strongly disagree"). Summary scores range from 0 to 15, higher scores indicate greater work strain.
Change in Caregiver Daily Psychological Distress | Day 1 to Day 8
  Using the daily version of the Non-Specific Psychological Distress Scale, each day, the caregiver will indicate how frequently they felt 14 negative/13 positive emotions over the past 24 hours on a 5-point scale from "none" to "all" of the time.

CONTACTS AND LOCATIONS:
Overall Officials: Karen A Roberto, PhD, Principal Investigator — Virginia Polytechnic Institute and State University; Jyoti Savla, PhD, Principal Investigator — Virginia Polytechnic Institute and State University
Locations (1):
- Virginia Polytechnic Institute and State University, Blacksburg, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
Not applicable; will not be sharing individual participant data with other researchers.

REFERENCES:
- See also: CareEx Study Website — https://careex.isce.vt.edu/